CLINICAL TRIAL: NCT03567122
Title: Attentional Focus Influence During Cranio-Cervical Flexion Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Francisco Xavier de Araujo, Pt, Principal Ivestigator, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MSS_ME_01
Record Dates: First submitted 2018-06-01; First posted 2018-06-25 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Neck; Anomaly; Muscle Weakness; Muscle Weakness Condition
Keywords: Cranio-cervical; Motor Control; Deep Flexor muscles
MeSH Terms: conditions — Congenital Abnormalities; Muscle Weakness

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Internal Focus of Attention (Experimental): 30 subjects will be randomized to this arm. Only internal focus of attention feedback instructions will be given during the execution and training performing the Cranio-Cervical Flexion Test. The subjects allocated to this arm will not be allowed to use the visual feedback traditionally provided during the Cranio-cervical Flexion Test.
  Interventions: Other: Internal Focus of Attention
- External Focus of Attention (Experimental): 30 subjects will be randomized to this arm. Only external focus of attention feedback instructions will be given during the execution and training performing the Cranio-Cervical Flexion Test. The subjects allocated to this arm will not be allowed to use the visual feedback traditionally provided during the Cranio-cervical Flexion Test. In addition, they will use just a laser point attached to the head to guide their cranio-cervical flexion.
  Interventions: Other: External Focus of Attention
- Control (Active Comparator): 30 subjects will be randomized to this arm. The participants allocated to this arm will be instructed as traditionally during the Cranio-Cervical Flexion Test. They will be given visual feedback while have their attention guided to the inner neck movement.
  Interventions: Other: Control

INTERVENTIONS:
Other: Internal Focus of Attention — Information already included in arm/group descriptions.
  Other Names: Internal Focus
  Arms: Internal Focus of Attention
Other: External Focus of Attention — Information already included in arm/group descriptions.
  Other Names: External Focus
  Arms: External Focus of Attention
Other: Control — Information already included in arm/group descriptions.
  Arms: Control

SUMMARY:
The purpose of this study is to termine if a different attentional focus would alter the motor control in cervical muscles during the cranio-cervical test.

DETAILED DESCRIPTION:
Asymptomatic subjects will be recruited to this study. Superficial electromyography of the Sternocleidomastoid, Range of Motion (ROM) and Cranio-Cervical Flexion Test (CCFT) will be measured before, immediately after change in focus of attention, 2 days after training under a particular focus of attention, and 7 days after training the task under the same focus of attention.

Subjects will be randomized into three groups: Internal focus of attention, external focus of attention and control group.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic subjects

Exclusion Criteria:

* Cervical pain
* Historic of trauma/surgery to the cervical or thoracic spine or upper limbs
* Temporomandibular pain
* Neurological or systemic disorder

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Electromyographic Activity of Sternocleidomastoid | Baseline, Immediately after baseline, Post-Training (2 days after the baseline), Retention (7 days after finished training)
  The Electromyography (EMG) signal amplitude will be determined by the root mean square (RMS) value computed over intervals of 1 s during each 10-s contraction. RMS will be expressed as a percentage of the maximum RMS value during the reference voluntary contraction.

SECONDARY OUTCOMES:
Cranio-cervical Range of Motion | Baseline, Immediately after baseline, Post-Training (2 days after the baseline), Retention (7 days after finished training)
  A neutral position and full range of active cranio-cervical flexion photograph will be taken using a digital camera. That camera will be positioned on a tripod horizontally parallel to the subject's head/neck region at a distance of 80 cm, anatomical markers positioned on the tragus of the ear, the mental protuberance of the mandible and the lateral aspect of the neck. Photos will be taken when the subject reached each level of the craniocervical flexion test. The Cranio-cervical Range of Motion will be expressed as relative percentage of degrees compared to the full range of motion.
Cranio-Cervical Flexion Test Performance | Baseline, Immediately after baseline, Post-Training (2 days after the baseline), Retention (7 days after finished training)
  Subjects will instructed to reach each one of the five stages (22-30 mmHg) of the test and hold the pressure as steady as possible for 10s. The stage will be mark as successful if the participant reaches the stage level and hold steady the pressure during the 10-s contrition. However, the individuals that reaches the stage-aimed pressure but are unable to maintain the pressure stable during the 10s contraction or use compensating strategies will be marked as unsuccessful.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Faria, PhD, PT, Study Director — Professor, Researcher
Locations (1):
- Universidade Federal de Ciências da Saúde, Porto Alegre, Rio Grande do Sul, Brazil